CLINICAL TRIAL: NCT01005108
Title: Acupuncture and Gabapentin for Hot Flashes Among Breast Cancer Survivors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UPCC 16108; NCI-2009-01315
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Hot Flashes
Keywords: Hot Flashes for Breast Cancer Patients
MeSH Terms: conditions — Hot Flashes | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- placebo pill (Experimental)
  Interventions: Drug: Gabapentin
- placebo accupuncture (Experimental)
  Interventions: Drug: Gabapentin
- accupuncture (Experimental)
  Interventions: Drug: Gabapentin
- gabapentin (Experimental)
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — Use of Gabapentin as a control intervention to evaluate the relative effects and adverse events of acupuncture for hot flashes

SUMMARY:
Overall Objectives: The overarching goal is to compare the effectiveness of acupuncture and gabapentin to their respective placebo controls in the treatment of hot flashes in breast cancer patients. The investigators primary specific aim will focus on determining the magnitude of response to placebo acupuncture versus placebo pills on hot flashes (HFs).

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 years or older with a history of Stage I, II or III breast cancer for at least 12 months.
2. Have been seen by an oncologist within the previous 6-month period and determined to be free of disease by clinical examination and history;
3. Experienced at least two hot flashes daily over the seven-day screening period as based on the Daily Hot Flash Diary.
4. Hot flashes have been present for at least a month before study entry.
5. Willing to use non-hormonal contraceptives during the duration of the study if patient is premenopausal.

Exclusion Criteria:

1. Having metastatic breast cancer ( IV)
2. Currently on chemotherapy or radiation therapy as adjuvant treatment
3. Started hormonal therapies such as tamoxifen or aromatase inhibitors within the last 4 weeks; or plan to change or terminate hormonal therapies in the next 14 weeks.
4. Started or changed with treatments for hot flashes, such as SSRIs or clonidine within the last 4 weeks; or plan to change or terminate these therapies in the next 14 weeks.
5. Current use of estrogen and/or progestin.
6. Pregnancy
7. Breast feeding
8. Bleeding disorder or current use of warfarin or heparin by patient history because of the use of needles.
9. Previous use of gabapentin for hot flashes.
10. Current use of any anti-convulsant.
11. Renal dysfunction defined as serum creatinine concentration above 1.25 times the upper limit of normal
12. Known allergy to gabapentin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2014-01-31 (Actual); Study Completion 2014-01-31 (Actual)

PRIMARY OUTCOMES:
Daily Hot Flash Diary (DHFD)-Primary Outcome (2 minutes per day) | Daily starting from baseline until week 12 and again for one week at week 24.

SECONDARY OUTCOMES:
Demographics -Covariates | 5 minutes
Hot Flash Related Daily Interference Scale (HFRDIS)-Secondary outcome | 3 minutes
Pittsburgh Sleep Quality Index (PSQI) - Secondary outcome | 6 minutes
Brief Fatigue Inventory (BFI) - Secondary Outcome | 3 minutes
HADS - Secondary Outcome | 2 minutes
Global Assessment Scale -Secondary Outcome | 30 seconds
Acupuncture Expectancy Scale (AES) - Secondary Aim | 1 minute
Creditability Rating of Acupuncture - Secondary Aim | 1 minute
Medication and CAM Usage -Covariates | 5 minutes
Actigraph Movement Measuring Device | 24 hrs/day for 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Jun J Mao, MD, MSCE, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the Unviersity of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Romero SAD, Li QS, Orlow I, Gonen M, Su HI, Mao JJ. Genetic predictors to acupuncture response for hot flashes: an exploratory study of breast cancer survivors. Menopause. 2020 Aug;27(8):913-917. doi: 10.1097/GME.0000000000001545. PMID 32217888
- [Derived] Garland SN, Xie SX, Li Q, Seluzicki C, Basal C, Mao JJ. Comparative effectiveness of electro-acupuncture versus gabapentin for sleep disturbances in breast cancer survivors with hot flashes: a randomized trial. Menopause. 2017 May;24(5):517-523. doi: 10.1097/GME.0000000000000779. PMID 27875389
- [Derived] Mao JJ, Bowman MA, Xie SX, Bruner D, DeMichele A, Farrar JT. Electroacupuncture Versus Gabapentin for Hot Flashes Among Breast Cancer Survivors: A Randomized Placebo-Controlled Trial. J Clin Oncol. 2015 Nov 1;33(31):3615-20. doi: 10.1200/JCO.2015.60.9412. Epub 2015 Aug 24. PMID 26304905